CLINICAL TRIAL: NCT06499844
Title: Comparing Approaches to Assess Nitric Oxide-dependent Cutaneous Vasodilation
Acronym: CAP NOVA
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202404816
Record Dates: First submitted 2024-06-26; First posted 2024-07-15 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Endothelial Function
MeSH Terms: interventions — Acetylcholine

STUDY DESIGN:
Intervention Model Description: All participants will complete one laboratory visit to assess endothelial function in the cutaneous microvasculature.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- assessment of microvascular endothelial function (Experimental): The investigators use intradermal microdialysis to deliver acetylcholine, L-NAME, and acetylcholine + L-NAME to the cutaneous microvasculature.
  Interventions: Drug: Acetylcholine

INTERVENTIONS:
Drug: Acetylcholine — acetylcholine, and acetylcholine + L-NAME (Nitric oxide synthase inhibitor) are locally and acutely delivered to the cutaneous microvasculature to assess endothelium- and nitric oxide-dependent dilation

SUMMARY:
The increase in skin blood flow in response to rapid local heating of the skin (i.e., cutaneous vasodilation) is commonly used to assess nitric oxide (NO)-dependent dilation and overall microvascular function. Historically, rapid local heating to 42°C was considered the standard approach for these assessments. More recently, many investigators have adopted rapid local to 39°C instead, based on its larger dependency on NO and therefore improved ability to quantify NO-dependent dilation without the use of pharmacological techniques. However, to date, only one direct methodological comparison between these protocols has been performed.

In this study, the investigators use the blood vessels in the skin as a representative vascular bed for examining mechanisms of microvascular dysfunction in humans. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) they examine the blood vessels in a nickel-sized area of the skin in young adults ages 18 - 30 years old. Local heating of the skin at the microdialysis sites is used to explore differences in mechanisms governing microvascular control. As a compliment to these measurements, the investigators also have participants fill out a variety of surveys to assess things such as sleep quality, physical activity, daily stressors, etc.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* 18-30 years of age

Exclusion Criteria:

* Current or recent (within 8 wks) use of medication that could conceivably alter microvascular function [including (but not limited to) stimulants, antihypertensives, HMG-CoA reductase inhibitors]
* Changes or alterations in medication status (starting a new, additional, or different medication or changing the dose of a current medication)
* Unstable or diagnosed chronic clinical disease, including cardiovascular, metabolic, renal, hepatic, autonomic, autoimmune, or dermatological disease (e.g., hypertension, heart disease, diabetes, hyperlipidemia, psoriasis)
* Body mass index <18.5 or >35 kg/m2
* Pregnancy (including a positive urine pregnancy test) or breast-feeding
* Known allergies to pharmacological agents or study drugs
* Non-English-speaking. Participants need to understand English to follow instructions and comply with procedures conducted during the screening and experimental visits.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Microvascular blood flow response to acetylcholine | baseline study visit (average of 4 hours)
  cutaneous vascular vasodilator response to exogenous acetylcholine perfusion; measured with laser-Doppler flowmetry coupled with intradermal microdialysis delivery of acetylcholine alone or co-infused with L-NAME
Microvascular blood flow response to local heat (42 degrees Celsius) | baseline study visit (average of 4 hours)
  cutaneous vascular vasodilator response to 42 degree local heat; measured with laser-Doppler flowmetry coupled with intradermal microdialysis delivery of lactated Ringer's, followed by L-NAME.
Microvascular blood flow response to local heat (39 degrees Celsius) | baseline study visit (average of 4 hours)
  cutaneous vascular vasodilator response to 39 degree local heat; measured with laser-Doppler flowmetry coupled with intradermal microdialysis delivery of lactated Ringer's, followed by L-NAME.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No